CLINICAL TRIAL: NCT05612451
Title: Outcome of Regenerative Endodontic Procedures for Necrotic Immature Permanent Teeth, Using Two Different Protocols: A Prospective Randomized Clinical Study.
Brief Title: Outcome of Regenerative Endodontic Procedures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: King Abdullah University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20180112
Record Dates: First submitted 2022-11-02; First posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Endodontic Disease
Keywords: Endodontic regeneration; Immature teeth; Randomized controlled trial
MeSH Terms: conditions — Dental Pulp Diseases

STUDY DESIGN:
Intervention Model Description: This randomized clinical trial aimed to assess and compare the clinical and radiographic outcomes of Regenerative Endodontic Procedures (REP) in treating non-vital immature permanent teeth using two intracanal medicaments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-setting calcium hydroxide (Experimental): Regenerative Endodontic Procedure utilizing non-setting calcium hydroxide as intracanal medicament
  Interventions: Procedure: Regenerative Endodontic Procedures; Other: non-setting calcium hydroxide
- modified triple antibiotic paste (Experimental): Regenerative Endodontic Procedure utilizing modified triple antibiotic paste as intracanal medicament
  Interventions: Procedure: Regenerative Endodontic Procedures; Other: modified triple antibiotic paste

INTERVENTIONS:
Procedure: Regenerative Endodontic Procedures — Regenerative Endodontic procedures were performed by one operator following similar protocols according to the clinical considerations for a regenerative procedure advised by the American Association of Endodontists and European Society of Endodontology
Other: non-setting calcium hydroxide — non-setting calcium hydroxide
  Arms: non-setting calcium hydroxide
Other: modified triple antibiotic paste — modified triple antibiotic paste
  Arms: modified triple antibiotic paste

SUMMARY:
Clinical management of immature non-vital (necrotic) permanent teeth is challenging, due to inherent structural weakness. Earlier management of such teeth relied on the traditional calcium hydroxide (Ca(OH)2) apexification procedure or the application of apical barriers However, neither procedure allows for promoting root dentin maturation. In 2004, a novel management technique for treating immature, non-vital teeth called regenerative endodontic procedures (REP; also known as revascularization) was introduced. This procedure allowed for continued root maturation presented in an increase in root length and dentin wall thickness. The key points of REP include minimal or no instrumentation of the dentinal walls, disinfection with irrigant solutions and intracanal medicaments, provocation of bleeding into the canal space for creation of a blood clot, capping with calcium silicate-based material, and an effective coronal seal to prevent reinfection of the root canal system. Several case reports and clinical studies reported promising results for REP treatment. However, studies widely varied in their treatment methods, hence the search for an optimal REP protocol is still ongoing. A recent review reported that the methodological quality of REP clinical trials available to date, was low with a moderate to high risk of bias. To date, only few studies evaluated the outcome of REPs based on different types of intracanal medicaments. These studies either presented a retrospective design, low sample size and/or short follow up period. Hence, the need for randomized, controlled clinical studies to provide persuasive evidence on the efficacy of different intracanal medicaments in REP is of utmost importance. The aim of this study is to prospectively assess and compare the clinical and radiographic outcomes of REP in non-vital immature permanent teeth using an intracanal medicament modified TAP or non-setting Ca(OH)2 paste. Forty-five patients yielding a total of 50 anterior and posterior non-vital immature teeth were randomly divided into 2 groups. REP utilizing either non-setting calcium hydroxide (Ca(OH)2) (n=25) or modified triple antibiotic paste (TAP) (n=25), as intracanal medicaments were performed. NeoMTA Plus was applied for coronal sealing. Cases were followed up clinically and radiographically for 24 months. Survival rate, success rate, and clinical outcome measures were analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Anterior or posterior tooth diagnosed with necrotic pulp (as a result of trauma, caries or anomaly) in the presence or absence of apical periodontitis.
2. an immature apex or open apex(an apical diameter wider than 1 mm and is radiographically visible)
3. Pulp space not needed for post and core restoration
4. A cooperative and Compliant patient/ parent
5. Patients not allergic to medicaments necessary to complete the procedure.

Exclusion Criteria:

1. medically compromised patient,
2. teeth with vertical fractures,
3. periodontally involved teeth,
4. non-restorable teeth,
5. teeth when bleeding could not be induced.

Ages: 7 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2024-06-27 (Estimated)

PRIMARY OUTCOMES:
treatment success | 36 months
  disappearance of clinical signs and symptoms including tenderness to percussion or palpation, a swelling or sinus tract, or spontaneous pain, and absence or reduction in the size of periapiacl radiolucency

SECONDARY OUTCOMES:
root elongation | 36 months
  increased root length
root maturation | 36 months
  increased root dentin thickness
root completion | 36 months
  apical closure

CONTACTS AND LOCATIONS:
Overall Officials: Aladdin A Al-Qudah, PhD, Principal Investigator — Jordan University of Science & Technology
Locations (1):
- Jordan University of Science & Technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting 12 months after publication
Access Criteria: will be sent by email, upon request

REFERENCES:
- [Result] Duggal M, Tong HJ, Al-Ansary M, Twati W, Day PF, Nazzal H. Interventions for the endodontic management of non-vital traumatised immature permanent anterior teeth in children and adolescents: a systematic review of the evidence and guidelines of the European Academy of Paediatric Dentistry. Eur Arch Paediatr Dent. 2017 Jun;18(3):139-151. doi: 10.1007/s40368-017-0289-5. Epub 2017 May 15. PMID 28508244
- [Result] Saoud TM, Zaazou A, Nabil A, Moussa S, Lin LM, Gibbs JL. Clinical and radiographic outcomes of traumatized immature permanent necrotic teeth after revascularization/revitalization therapy. J Endod. 2014 Dec;40(12):1946-52. doi: 10.1016/j.joen.2014.08.023. Epub 2014 Oct 16. PMID 25443280
- [Result] European Society of Endodontology (ESE) developed by:; Krastl G, Weiger R, Filippi A, Van Waes H, Ebeleseder K, Ree M, Connert T, Widbiller M, Tjaderhane L, Dummer PMH, Galler K. European Society of Endodontology position statement: endodontic management of traumatized permanent teeth. Int Endod J. 2021 Sep;54(9):1473-1481. doi: 10.1111/iej.13543. Epub 2021 Jun 20. PMID 33934366
- [Result] Sponchiado-Junior EC, Vieira WA, Frozoni M, Herkrath FJ, de-Jesus-Soares A. CONSORT Compliance in Randomized Clinical Trials of Regenerative Endodontic Treatments of Necrotic Immature Teeth: A Scoping Review. J Endod. 2021 Nov;47(11):1751-1766. doi: 10.1016/j.joen.2021.07.017. Epub 2021 Aug 3. PMID 34352304
- [Result] Chan EK, Desmeules M, Cielecki M, Dabbagh B, Ferraz Dos Santos B. Longitudinal Cohort Study of Regenerative Endodontic Treatment for Immature Necrotic Permanent Teeth. J Endod. 2017 Mar;43(3):395-400. doi: 10.1016/j.joen.2016.10.035. Epub 2017 Jan 19. PMID 28110920
- [Result] ElSheshtawy AS, Nazzal H, El Shahawy OI, El Baz AA, Ismail SM, Kang J, Ezzat KM. The effect of platelet-rich plasma as a scaffold in regeneration/revitalization endodontics of immature permanent teeth assessed using 2-dimensional radiographs and cone beam computed tomography: a randomized controlled trial. Int Endod J. 2020 Jul;53(7):905-921. doi: 10.1111/iej.13303. Epub 2020 Apr 30. PMID 32249441